CLINICAL TRIAL: NCT05422404
Title: Comparison of Anti-Reflux Mucosal Ablation(ARMA) With Anti- Reflux Mucosectomy(ARMS) in Treatment of Gastroesophageal Reflux Disease- A Randomized Controlled Trial
Brief Title: Anti-Reflux Mucosal Ablation(ARMA) and Anti-Reflux Mucosectomy(ARMS) in Gastroesophageal Reflux Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-02-003C
Record Dates: First submitted 2022-05-19; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Gastroesophageal Reflux Disease; Endoscopy
Keywords: Anti-Reflux Mucosal Ablation; Gastroesophageal Reflux Disease; Endoscopic intervention; Anti- Reflux Mucosectomy
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic GERD patient reciving Anti-Reflux Mucosal Ablation (Experimental): 150 chronic GERD patients will be enrolled from our outpatient clinic. The inclusion criteria are as following: 20-75 years of age, history of GERD over 1 year, who had received daily PPIs or H2 antagonists over 6 month for GERD treatment, and having persistent typical GERD symptoms (acid reflux sensation or heartburn) or atypical GERD symptoms (hoarseness, cough, acid related chest pain, laryngitis) when off PPI or H2 antagonists therapy, defective gastroesophageal Defective junction reciving Anti-Reflux Mucosal Ablation.
  Interventions: Procedure: Anti-reflux mucosal ablation
- Chronic GERD patient reciving Anti-Reflux Mucosectomy (Active Comparator): 150 chronic GERD patients will be enrolled from our outpatient clinic. The inclusion criteria are as following: 20-75 years of age, history of GERD over 1 year, who had received daily PPIs or H2 antagonists over 6 month for GERD treatment, and having persistent typical GERD symptoms (acid reflux sensation or heartburn) or atypical GERD symptoms (hoarseness, cough, acid related chest pain, laryngitis) when off PPI or H2 antagonists therapy, defective gastroesophageal Defective junction reciving Anti-Reflux Mucosectomy
  Interventions: Procedure: Anti-Reflux Mucosectomy

INTERVENTIONS:
Procedure: Anti-Reflux Mucosectomy — ARMS will be performed using gastroscope . The preparation and endoscopy procedure will be done as in regular practice with conscious sedation. The upper gastrointestinal tract will be evaluated in detail first. Then Endoscopic mucosal resection(EMR) will performed at E-C junction, gastric cardia side. About 50%-70% of the EGJ circumference will be resected to create artificial ulcer which will lead to mucosal contraction during the healing process.
  Arms: Chronic GERD patient reciving Anti-Reflux Mucosectomy
Procedure: Anti-reflux mucosal ablation — ARMA will be performed using gastroscope . The preparation and endoscopy procedure will be done as in regular practice with conscious sedation. Mucosal ablation will be performed in retroflex fashion following. Then APC with soft coagulation(effect 2, 40W) will be used to mark the area that not going to be ablated at gastric carida over the great curvature direction, about 1.5 scope width. Then submucosa injection with saline and indigo carmine dye will be performed using a 25 guage needle.
  Arms: Chronic GERD patient reciving Anti-Reflux Mucosal Ablation

SUMMARY:
According to the current published data and treatment mechanism, ARMS may led to more stenosis while ARMA may be less effective in long term follow-up. The changes of patient's life quality , UGI tract microbiota before and after different endoscopic treatment are also limited. So we want to conduct a exploratory prospective randomized controlled study in evaluating the mucosal healing, demand of PPI, life quality, emotion status, sleep quality, esophageal motility/ acid exposure and saliva microbiota between chronic GERD patients receiving ARMS and ARMA treatment.

DETAILED DESCRIPTION:
In this study, we will enroll 150 patients with chronic GERD. Estimated 40% of patients will be excluded from the inclusion and exclusion criteria. Of 90 patients eligible for the study, estimating 20% may drop out before receiving ARMS or ARMA. Estimated 72 patients will be randomized to receive ARMS or ARMA for GERD treatment. After ARMA, all patients will receive 4 weeks of PPI treatment. Endoscopy and questionnaire follow-up will be performed on week 2, 2 months, 6 months and 12 months after treatment while HRM and 24 hours pH impedance study will be performed 6 months after treatment.

The study will be carried out in 4 years. In the 1st to 3rd year of study, estimating 60,60,30 patients will be evaluated and entered the study in the 1st, 2nd and fisr half of 3rd year. Then all the patients will be followed until the first half of 4th year. At the second half of the 4th year, the saliva sample will be processed, data will be analyzed, and the result will be written.

1. st year study:60 patients enrollment, evluation and receiving endoscopy treatment with follow-up
2. nd year study:60 patients enrollment, evluation and receiving endoscopy treatment with follow-up
3. rd year study:30 patients enrollment, evluation and receiving endoscopy treatment with follow-up
4. th year study: complete all patients follow-up, sample processing, data analysis and report writing

ELIGIBILITY:
Inclusion Criteria:

* 20-75 years of age,
* History of GERD over 1 year

Exclusion Criteria:

* body mass index (BMI) > 35
* Hiatal hernia > 2cm
* Esophageal ulcer
* Esophageal stricture
* Barrett's esophagus (Prague criteria: C>1cm, M>=2cm)
* Major esophageal motility disorders
* Gastroparesis
* Pregnancy or plans for pregnancy in the next 12 months
* Immunosuppressive therapy
* Cirrhosis
* Portal hypertension and/or varices
* Previous gastric or esophageal surgery
* Esophageal diverticulum
* Scleroderma or dermatomyositis
* Coagulation disorders
* Anti-platelet or anticoagulants use

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Reflux synptom improvement after different treatment. | 6 months
  Reflux synptom improvement in 6 months after ARMS and ARMA. Complete remission group will be defined as GERD-Q score of <8 and discontinuing PPI medication. Patients with post- ARMS GERD-Q score of <8 and reduced PPI medication will be allocated to the partial response group. Others will be defined as non-response group.

SECONDARY OUTCOMES:
Comparisons of GERD DeMeester scores | 12 months
  DeMeester scores using 24 hours PH monitor for comparison of ARMS and ARMA groups.
Comparisons of GERD acid exposure time | 12 months
  Acid exposure time using 24 hours PH monitor for comparison of ARMS and ARMA groups.
improvement of GERD-Health Related Quality of Life Questionnaire (GERD-HRQL) | 6 months
  improvement ofGERD-Health Related Quality of Life Questionnaire (GERD-HRQL) 6 months after ARMS or ARMA procedure.
change of saliva microbiota | 2 months
  change of saliva microbiota before and after ARMS or ARMA procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Yen po Wang, Study Director — Taipei veteran general hospital

REFERENCES:
- [Background] Eusebi LH, Ratnakumaran R, Yuan Y, Solaymani-Dodaran M, Bazzoli F, Ford AC. Global prevalence of, and risk factors for, gastro-oesophageal reflux symptoms: a meta-analysis. Gut. 2018 Mar;67(3):430-440. doi: 10.1136/gutjnl-2016-313589. Epub 2017 Feb 23. PMID 28232473
- [Background] Chen TS, Chang FY. The prevalence and risk factors of reflux esophagitis among adult Chinese population in Taiwan. J Clin Gastroenterol. 2007 Oct;41(9):819-22. doi: 10.1097/01.mcg.0000225658.30803.79. PMID 17881927
- [Background] Hung LJ, Hsu PI, Yang CY, Wang EM, Lai KH. Prevalence of gastroesophageal reflux disease in a general population in Taiwan. J Gastroenterol Hepatol. 2011 Jul;26(7):1164-8. doi: 10.1111/j.1440-1746.2011.06750.x. PMID 21517967